CLINICAL TRIAL: NCT07012824
Title: Couple-Based Crisis Response Planning for Veterans
Brief Title: Couple-Based Crisis Safety Planning
Acronym: CRP-C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Bauer, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROJECT00009562; HT94252410658 (Other Grant/Funding Number: Assistant Secretary of Defense for Health Affairs endorsed by the Department of Defense)
Record Dates: First submitted 2025-05-08; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideas; Suicidal Ideation; Crisis; Emotional; Suicide Attempts; Suicidal and Self-injurious Behaviour; Suicidal Impulses
Keywords: Veteran safety; Suicide risk; Crisis safety plan; Suicide crisis; intervention
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two conditions: (1) CRP (control) where a Veteran will undergo the traditional CRP intervention, without the help participation of a romantic partner, and (2) CRC-P, where couples with at least one Veteran in the relationship will work together to complete the CRP-C intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Crisis Response Planning (Active Comparator): This arm will utilize the traditional Crisis Response Plan protocol. This arm will not utilize the help of a romantic partner in creating a crisis safety plan for the participating Veteran.
  Interventions: Behavioral: Crisis Response Planning
- Couples-based Crisis Response Planning (Experimental): This arm will utilize Couples-based Crisis Response Planning. This method of intervention involves the participation of the romantic partner of a Veteran who is receiving the intervention.
  Interventions: Behavioral: Couples-based Crisis Response Planning

INTERVENTIONS:
Behavioral: Crisis Response Planning — Crisis Response Planning (CRP) is a brief, one-time intervention that teaches individuals to notice warning signs of an impending crisis (e.g., suicidal crisis) and provide them with skills to help reduce suicide risk.
  Other Names: Safety Planning; CRP
  Arms: Traditional Crisis Response Planning
Behavioral: Couples-based Crisis Response Planning — This intervention expands on traditional CRP by integrating the intimate partner into the intervention. Among service members, intimate partners are the group most likely to be told about suicidal thoughts prior to a suicide attempt.
  Other Names: CRP-C
  Arms: Couples-based Crisis Response Planning

SUMMARY:
Suicide is a leading cause of death in Veterans. Suicide rates among Veterans have increased approximately 36% from 2001 to 2020. Veterans are at increased risk for suicide compared to non-Veterans, with the rate of suicide death being 57.3% higher for Veterans than non-Veterans. The present study will pilot test a virtual couple-based crisis response plan (CRP-C) for Veterans in order to reduce crisis symptoms and decrease suicide risk.

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial of a novel, virtually-delivered, single- session Couple-Based Crisis Response Plan (CRP-C) to reduce suicide crisis symptoms and decrease suicide risk in a community-based Veteran sample in Georgia. Crisis response planning (CRP; also referred to as "Safety Planning") is a brief, one-time intervention that teaches individuals to notice warning signs of an impending crisis (e.g., suicidal crisis) and provide them with skills to help reduce suicide risk. CRP has been shown to be effective at reducing suicidal behaviors. A strong line of research shows that a relationship with an intimate partner (e.g., a spouse) is often a major protective factor for preventing suicide risk. Further, partners are often the only (and last) people Veterans talk about suicidal thoughts with. Despite this, clinicians do not have any brief interventions (like CRP) that leverage the partner relationship to make the intervention more effective. In addition, past work has heavily focused on providing CRP to Veterans who have disclosed suicide risk. However, investigators know that many Veterans do not disclose risk at all and do not seek out treatment for suicidal thoughts because of stigma. It may be more beneficial to give CRP to Veterans who exhibit less-stigmatized symptoms that are strongly associated with suicide risk (e.g., sharp increases in agitation, insomnia, irritability, etc.) but who may not yet have developed suicidal ideation or are unwilling to disclose suicidal ideation. This approach may provide more Veterans and their partners with the skills needed to navigate a suicidal crisis and prevent suicide attempts/deaths.

This project will test the efficacy of a virtually-delivered, single-session Couple-Based Crisis Response Plan (CRP-C) in decreasing suicide crisis symptoms in a community-based Veteran sample compared to standard (individual) Crisis Response Planning (CRP). The investigators will enroll 50 couples where at least one of the partners is a Veteran. Couples will be randomized to receive traditional CRP or CRP-C via a virtual, one-time session. The CRP-C is comprised of the same components as traditional CRP, but with several key additions: 1) The partner also completes the CRP-C on behalf of the Veteran; 2) CRP-C contains an additional section that includes practical steps for broaching crisis-related conversations with the partner (i.e., helpful/unhelpful language, helpful/unhelpful actions, alterations for severe crises); 3) After completing the CRP-C independently, the Veteran and partner compare responses to increase awareness for both parties and allow the partner to offer additional suggestions and ask clarifying questions. Veterans will be surveyed 3x per day for thirty days to assess fluctuations of crisis symptoms and suicide risk, and complete a 3-month follow-up assessment. The investigators will test two advertisements (recruiting for crisis symptoms, recruiting for suicide risk) for the same study to test recruitment strategy effects on recruitment outcomes.

Our main aims are to:

1. Investigate the acceptability and feasibility of CRP-C
2. Test the effects of CRP-C on reducing crisis symptoms
3. Examine the effect of recruitment strategies on recruitment rates.

To achieve the study's primary aim (gather feasibility and acceptability data), the investigators chose a two-arm, repeated measures approach to quantitatively examine the intervention.The investigators will compare feasibility and acceptability with traditional CRP, as CRP is the current standard of care for the VA, medical centers, and many outpatient clinics for patients at increased risk for suicide. Given that CRP-C is ultimately meant to decrease STBs, it is critical to examine if adverse events and tolerability are similar in the two approaches to ensure safety of future participants and their partners. Due to the highly dynamic nature of suicidal crises, STBs, and STB risk factors, the investigators will use EMA methodology for higher temporal resolution to help understand potential effects of CRP-C.

Given the difficulty of engaging Veterans with suicide prevention interventions, the investigators will also test if recruiting based on non-stigmatized crisis symptoms leads to increased enrollment compared to recruiting to reduce STBs. Throughout, the investigators will also use qualitative methods to obtain a deeper understanding of how to tailor the intervention to couples in the Veteran population and help identify contextual aspects implementing the CRP-C that will not be measured during the pilot but would be assessed in the subsequent trial. Qualitative feedback will also help guide interpretation and application of the quantitative findings and provide additional information on intervention fidelity.

Specific Aim 1: Gather feasibility and acceptability data

Specific Aim 2: Use EMA methodology for higher temporal resolution to help understand potential effects of CRP-C

Specific Aim 3: Test if recruiting based on non-stigmatized crisis symptoms leads to increased enrollment compared to recruiting to reduce suicidal thoughts and behaviors

ELIGIBILITY:
Inclusion Criteria:

* (At least) One participant from the couple must have Veteran status
* Currently resides in Georgia
* English speaking
* The Veteran must own a smartphone
* Veteran must have experienced crisis symptoms in the past three months. At least 1 symptom of entrapment, and at least 1 symptom from 2 of the associated disturbance categories [i.e. affective disturbance, loss of cognitive control, hyperarousal, or social withdrawal]
* Currently be in a committed relationship for at least one year
* The Veteran must be able to present a copy of DD form 214 (Certificate of Release or Discharge from Active Duty issued by the U.S. Department of Defense)

Exclusion Criteria:

* Non-English speaking
* Under 18 years of age
* Resides in a different state than Georgia
* Either partner reports injury or fear resulting from intimate partner violence in the past three months.
* Participants who meet study criteria for imminent suicide risk Depressive Symptom Index - Suicidality Subscale (Joiner et al., 2002), defined as a DSI- SS score of 7 or greater, or selecting "3" on items B [formulated plan] or D [constant urge to kill self (I. H. Stanley et al., 2021)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Measured at 3-month follow-up appointment (Post-intervention)
  Higher scores indicate greater acceptability of the present intervention. The minimum score is 4 and the maximum possible score is 20.
Feasibility Measure of Intervention (FIM) | Measured at 3-month follow-up appointment (Post-intervention)
  Higher scores indicate greater feasibility of the present intervention. The minimum score is 4 and the maximum possible score is 20.
Intervention Appropriateness Measure (IAM) | Measured at 3-month follow-up appointment (Post-intervention)
  Higher scores indicate greater appropriateness of the present intervention. The minimum possible score is 4 and the maximum possible score is 20.
Suicide Crisis Inventory-2 | Measured during eligibility screening, baseline and at 3-month follow-up
  Suicide crisis symptoms will be assessed using a short form version of the Suicide Crisis Inventory - 2 (SCI-2) during eligibility screener. The SCI-2-SF is a 9-item self-report measure that assesses crisis symptoms over the past several days across five subscales: 1) Entrapment; 2) Affective Disturbance; 3) Loss of Cognitive Control; 4) Hyperarousal; and 5) Social Withdrawal, with selected items recorded such that higher scores are indicative of more severe SCS symptoms. The full 61-item measure will be utilized in later stages of data collection (i.e. baseline assessment and 3-month follow-up assessment). The maximum total score for the short form version is 36. The maximum total score for the standard 61-item version of the measure is 244. Minimum possible scores for both versions of the scale are 0.
Recruitment Engagement | Monitored throughout enrollment phase (i.e. from start of enrollment until participant quota is met). This will occur over approximately a 3-month time frame. This data will be analyzed along with other outcomes after data collection has concluded.
  Once the desired participant quota (50 couples) is met, the study team will analyze the means by which participants were recruited. This study utilizes two different advertisements that describe the same study, but with different language. The study team will assess which type of advertisement yielded more engagement, once all participants are enrolled.

SECONDARY OUTCOMES:
The Couples Satisfaction Index (CSI) | Measured at baseline and at 3-month follow-up
  Relationship quality will be assessed using the Couples Satisfaction Index. The CSI is a widely-used and well-validated 32-item self-report measure that assesses relationship quality, and has been used for psychosocial interventions for military couples. Higher scores indicate greater satisfaction with one's relationship. The maximum total score for this scale is 161. The minimum possible score is 0.
Difficulties in Emotion Regulation Scale (DERS) | Measured at baseline and at 3-month follow-up
  Emotion regulation will be assessed using the Difficulties in Emotion Regulation Scale. The DERS is a widely-used 36-item self-report measure that assesses emotion dysregulation and six subfactors: 1) Awareness; 2) Clarity; 3) Goals; 4) Impulse; 5) Non-Acceptance; and 6) Strategies. The measure is well-validated and has been used extensively in Veteran and military samples. Higher scores suggest greater problems with emotion regulation. The maximum possible total score is 180. The minimum possible total score is 36.
Cognitive Flexibility Inventory (CFI) | Measured at baseline and at 3-month follow-up
  Cognitive flexibility will be assessed using the Cognitive Flexibility Inventory. The CFI is a well-validated 20-item self-report measure that measures three aspects of cognitive flexibility: 1) Controllability Perception; 2) Alternative Explanation Awareness; and 3) Alternative Solution Generation. The maximum possible score on this scale is 140, and the minimum possible score is 20, with higher scores indicating greater cognitive flexibility.
Theory of Planned Behavior Questionnaire (TPBQ) | Measured at baseline and at 3-month follow-up
  Behavioral intention will be assessed using a Theory of Planned Behavior Questionnaire (TPBQ). The TPBQ is a 9-item version of the scale that was developed using the guidelines set forth by Ajzen (2006) and measures: 1) Attitude Toward Behavior; 2) Injunctive and Descriptive Norms; 3) Perceived Behavioral Control; 4) Intention; and 5) Past Behaviors. The scale was modified to fit the scope of the intervention that takes place in the study (i.e. Crisis Response Planning) This scale is scored in 5 different dimensions with a maximum total score of 63 and a minimum possible total score of 9.
Center for Epidemiologic Studies Depression Scale (CES-D) | Measured at baseline and at 3-month follow-up
  A self-report depression scale for research in the general population. Scores range from 0-60. A score equal to or above 16 indicates a person at risk for clinical depression.
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Administered one time during a 3-hour intervention session
  The Diagnostic Interview for Anxiety, Mood, and ObsessiveCompulsive and Related Neuropsychiatric Disorders will be used to assess current and lifetime histories of mental disorders to characterize the sample. This is necessary to understand the clinical severity of our sample in relation to previous CRP studies to guide interpretations for generalizability. The DIAMOND is a well-validated and widely-used semi-structured interview designed to assess for DSM-5 diagnoses. Screener questions and follow-up modules will be administered for the following disorders: Social Anxiety Disorder, Panic Disorder, Agoraphobia, Generalized Anxiety Disorder, Persistent Depressive Disorder, Major Depressive Disorder, Bipolar I & II Disorders, Obsessive-Compulsive Disorders, Acute Stress Disorder, Post-traumatic Stress Disorder, Adjustment Disorder, Substance Use Disorder, and Attention Deficit/Hyperactivity Disorder.
Columbia Suicide Severity Rating Scale (CSSRS) | Measured one time during a 3-hour intervention session
  This protocol includes two subscales from the Screening version of the Columbia-Suicide Severity Rating Scale © (C-SSRS): Severity of Suicidal Ideation and Suicidal Behavior. Both subscales provide definitions of suicidal ideation and behavior and corresponding probes. The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal, self-injurious behavior.
  The Current version of the C-SSRS assesses suicidality during a two time periods-ideation in the past month and suicidal behavior in the past 3 months.
Patient Health Questionnaire (PHQ-9) | Measured at baseline and at 3-month follow-up
  Depressive symptoms will be measured by the Patient Health Questionnaire-9. The PHQ-9 is a widely used 9- item self-report measure that assesses depressive symptoms over the past two weeks. The maximum possible score is 27 and the minimum possible total score is 0, with higher scores indicating greater severity of depressive symptoms.
Generalized Anxiety Disorder Screener (GAD-7) | Measured at baseline and at 3-month follow-up
  Anxiety symptoms will be measured by the Generalized Anxiety Disorder - 7. The GAD-7 is a widely used 7-item self-report measure that asses anxious symptoms over the previous two weeks. The maximum possible score is 21 and the minimum possible total score is 0, with higher scores indicating greater severity of anxiety symptoms
Disability Assessment (WHODAS 2.0) | Measured at baseline and at 3-month follow-up
  The investigators will use the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) to assess health and disability. The WHODAS 2.0 is a 12-question self-report measure that covers six domains: 1) Cognition; 2) Mobility; 3) Self-care; 4) Getting Along; 5) Life Activities; and 6) Participation. The maximum possible converted summary score is 100 and the minimum score is 0, with higher scores indicating a greater level of disability.
DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure-Adult | Measured at baseline and at 3-month follow-up
  Assesses mental health domains across several psychiatric diagnoses. This measure consists of 23 questions and assesses 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. Items ask individuals to rate how often they are bothered by symptoms in the last two weeks. A rating of mild (i.e., 2) or greater on any item within a domain (except for substance use, suicidal ideation, and psychosis) may serve as a guide for additional inquiry and follow up to determine if a more detailed assessment for that domain is necessary. For substance use, suicidal ideation, and psychosis, a rating of slight (i.e., 1) or greater on any item within the domain may serve as a guide for additional inquiry and follow-up to determine if a more detailed assessment is needed.

OTHER OUTCOMES:
Suicide Crisis Symptoms (SCS-2) | Measured 3 times a day for 30 days after intervention session
  Suicide crisis symptoms will be measured using an abbreviated version of the SCS-2. Two to three items exhibiting the largest factor loadings for each of the five subfactors were extracted, resulting in 17 items. These items were then edited to be in the present tense ("Please indicate how you are feeling on the following items") and replaced with a visual analogue scale (0-100), which is similar to past EMA studies assessing suicide risk and associated variables. Higher scores indicate greater severity of crisis symptoms.
Suicide Risk Assessment (DSI-SS) | Measured 3 times a day for 30 days after intervention session
  Suicide risk will be assessed using the Depressive Symptom Index - Suicide Subscale (DSI-SS). This is a 4-item self-report measure that assesses current risk. Higher scores indicate greater levels of risk. The maximum possible total score for this scale is 12 and the minimum possible total score is 0
Crisis Response Planning Engagement | Measured 3 times a day for 30 days after intervention session
  Crisis response planning engagement will be assessed using nine binary ("Yes/No") self-report items to understand if participants did any of the following since their last survey: 1) Identify warning signs; 2) Internal coping strategies; 3) Activity based distractions; 4) Social distractions; 5) Location change; 6) Discuss thoughts with partner or others; 7) Contacted professionals; 8) Hospitalization; and 9) Lethal means safety. Higher scores indicate greater level of engagement with the current intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian W. Bauer, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be submitted to the National Institute of Mental Health (NIMH) Data Archive (NDA) at the National Institutes of Health (NIH)
Supporting Information: ICF